CLINICAL TRIAL: NCT05223348
Title: Examining the Role of Perceived Body Boundaries and Spatial Frame of Reference in the Mechanism of Action of a Body Scan Meditation in Reducing Emotional Eating: A Randomized Controlled Study
Brief Title: Examining the Role of Perceived Body Boundaries and Spatial Frame of Reference in the Effect of a Mindfulness Meditation in Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: McGillU
Record Dates: First submitted 2021-12-16; First posted 2022-02-03 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly assigned to either the experimental condition, a body scan meditation, or a control condition, a listening task, using a random digit generator. This randomization will be done in a way that is blinded from the participants to ensure that knowledge of the practice to which they are assigned does not impact how they respond to the self-report questionnaires. In addition, the researcher guiding the mood induction will also remain blind to the participant allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Scan Meditation (Experimental): The experimental condition involves participants listening to a 16-minute recording of a body scan meditation. The body scan condition guides participants to focus on their bodily sensations separately, then together as a whole.
  Interventions: Other: Meditation practice
- Listening Task (Active Comparator): The active comparer condition involves participants listening to a 16-minute recording of text that describes the human musculoskeletal system. The text will be narrated by a female voice to match the body scan meditation. In addition, the focus on the body in the text of the active condition matches the focus on the body in the body scan meditation and, as such, controls for demand characteristics.
  Interventions: Other: Meditation practice

INTERVENTIONS:
Other: Meditation practice — Our intervention will involve two meditation exercises. 1) the experimental condition (body scan meditation). 2) the active comparator condition (listening task)

SUMMARY:
Emotional eating, or overeating in response to emotions, is problematic because of its link to weight gain, obesity, and psychopathology such as bulimia and binge eating disorder. To date, a vast amount of research has studied the psychological processes that cause individuals to overeat in response to emotions in an effort to develop ways to help individuals reduce their emotional eating. The aim of the current project is to study two psychological processes that can potentially be positively influenced to improve well-being: perceived body boundaries and a person's spatial frame of reference. Particularly, the investigators will examine how perceived body boundaries and spatial frames of reference can be positively influenced through a body scan meditation and thereby improve emotional eating. Perceived body boundaries refers to the continuum along which the self is experienced, from a body-encapsulated entity that is separate from the surrounding world to a more diffuse entity that is more connected with others and the environment. Spatial frames of reference describes the region within one's perception, often based in the body and construed as the self, that may be experienced as egocentric, through a preoccupation with internal events, or as allocentric, with feelings of unity and interdependence with others and the environment. One way for individuals to experience more diffuse body boundaries and allocentric frames of reference is through a body scan meditation. In this practice, individuals are instructed to intentionally shift their attention to various parts of the body and to notice what happens without judging or reacting. Thoughts and emotions are briefly noted if they arise, and attention is shifted back to the body. Recent research has shown that when individuals practice the body scan meditation, individuals are likely to experience greater positive emotions, lower negative emotions, lower ruminations, and higher psychological wellbeing. In addition, research has shown that individuals are able to experience more diffuse perceived body boundaries and more allocentric frames of reference through a body scan meditation. Based on this work, the researchers predict that when emotional eaters practice the body scan meditation, emotional eaters will experience more diffuse body boundaries, more allocentric frames of reference, and lower ruminations, which could in turn reduce their negative affect and food cravings. The researchers will test this hypothesis by asking emotional eaters to complete questionnaires that measure perceived body boundaries, spatial frames of reference, ruminations, negative emotions, and food cravings before and after a body scan meditation. To ensure that any changes in these measures are due to the meditation, the researchers will compare these findings with emotional eaters who complete the same measures before and after a control listening task. The findings of the current study will be used to recommend the body scan meditation to support emotional eaters in regulating their emotions, cravings, and eating behaviors.

DETAILED DESCRIPTION:
Emotional eating, or overeating in response to negative emotions is problematic because the overconsumption of high-caloric and high-fat foods can result in weight gain and obesity. It has also been linked to binge eating in bulimia nervosa and binge eating disorder.

Thus far, research examining the processes underlying emotional eating has used a number of different methods including self-report questionnaires, laboratory studies, and testing in naturalistic settings. Recently, our team used qualitative methodology to understand the phenomenology, or first-person subjective experience, of individuals while emotionally eating. The investigators interviewed eight individuals who emotionally ate and collected 16 hours of interview data using explicitaiton interviews, a type of interviewing method developed by Pierre Vermersch that aims to access an individual's phenomenology of an event by guiding them to relive the event in the present moment through a body-centered perspective. Preliminary thematic analysis of the data showed that most of the individuals described a theme of "thinking a lot" in response to negative emotions that they experienced. This is in line with a narrative focus that involves linking subjective experiences through time using thoughts of self-traits, traits of others, memories of the past, and aspirations of the future. In response to this narrative mode of functioning, individuals then described themes of "looking forward to the sensory experience" of food and consequently "enjoying the sensory experience," "not thinking about my stressors," and "being in the moment" while eating. This shift to sensory experience is in line with an experiential focus that involves inhibition of cognitive elaboration in favor of attending to present-moment sensory objects, including feelings and sensations rooted in the body.

The two modes of self-focus seen in our qualitative study of the phenomenology of emotional eating map on to modes of psychological functioning at the level of the self as described by, which can be used to understand how self-related processes impact emotional eating in order to help individuals reduce this behavior. Specifically, the theme of "thinking a lot" or rumination seen in our qualitative study can be mapped onto what Gallagher describes as the narrative self, characterized by mental activities such as thoughts, emotions, and motivations, linked to one's past and future. In this state of functioning, mental contents are experienced in a way that is identified with one's self, called experiential fusion or cognitive fusion, which leads to the perception of being the one who is thinking the thoughts or experiencing the emotions. While such a perception is adaptive for cognitive and social functioning (such as through a central locus of control, sense of identity, etc), an overemphasis on the sense of self, particularly when it is negative, is maladaptive. For example, narrative self-functioning that is high in rumination, negative self-judgments, cognitive fusion, and mind-wandering has been linked to a variety of psychopathologies, such as anxiety and depression. On the other hand, themes of "being in the moment", "enjoying the sensory experience," etc. seen in our qualitative study can be mapped onto what Gallagher describes as the minimal self, also referred to as the embodied self, because it consists of basic or core processes that are phenomenologically related to the body, such as sensorimotor experiences, sense of agency, and sense of ownership. In addition, the minimal self, dependent on sensory processing, is thought to allow for the parsing of "self" from "not-self" through body-based processes, such as shifts in perceived body boundaries and spatial frames of reference. Specifically, perceived body boundaries describe the degree to which the self is experienced as a discrete, body-encapsulated entity, separate and isolated from the surrounding world. Thus, when one perceives their body boundaries as more salient, a greater sense of separation of oneself from others and the environment is experienced. When one's body boundaries are perceived as more diffuse, higher levels of happiness are experienced. Similarly, the spatial frame of reference describes the region within one's perception, often based in the body and construed as the self, that is involved in the sense of connection between self, others, and the environment. Particularly, one's spatial frame of reference may be experienced as egocentric, or through a self-centered preoccupation with internal, private events, constraining the sense of self within the physical body's boundary, or allocentric, through distributed feelings of unity and interdependence with the others and the environment. More diffuse body boundaries and more allocentric frames of reference have been found to be associated with greater compassion for self and others, altruism, and psychological wellbeing.

One way to engage with the minimal self and increase wellbeing outcomes without relying on eating is through the practice of mindfulness, described as "paying attention in a particular way: on purpose, in the present moment, and non-judgmentally." For example, during the body scan meditation, a type of mindfulness practice, individuals are instructed to intentionally shift their attention to various parts of the body and to notice what happens without judging or reacting. If thoughts and emotions arise, they are briefly noted, and attention is shifted back to the body. This attention training facilitated a shift of attention from a thought-based narrative focus to sensory-based interoceptive awareness through cognitive defusion, or the ability to gain psychological distance from thoughts and feelings by seeing them as mere events in the mind, and equanimity, or an even-minded mental disposition towards all objects of experience regardless of their affective valence or source. As such, by practicing a body scan meditation, individuals are able to reduce focus on self-specifying cognitive processes that differentiate the self from not-self and experience more diffuse perceived body boundaries and more allocentric frame of reference, which lead to increased positive emotions and decreased negative emotions. Recent research has investigated the influence of the mindfulness meditation on emotions, perceived body boundaries, and spatial frames of reference. For example, Dambrun studied the effect of a body scan mindfulness meditation on happiness and anxiety and found a greater reduction in the salience of perceived body boundaries in the body scan condition compared to the control condition. Furthermore, he found that the change in perceived body boundaries was accompanied by an increase in happiness and decrease in anxiety and that the change in happiness was mediated by the change in perceived body boundaries. Similarly, a study by Hanley and Garland showed that a brief mindfulness practice encouraged more allocentric frames of reference and that more allocentric frames mediated the effect of mindfulness induction on affective state by increasing positive affect and decreasing negative affect. Finally, Hanley found that five sessions of mindfulness meditation training decreased perceived body boundaries and encouraged more allocentric frames of reference and that the effect of mindfulness training on allocentric frames of reference was mediated by decreased perceived body boundaries.

Within emotional eating, negative emotions lead to overeating through food cravings and an inability to down-regulate them. A food craving is defined as an intensely strong desire for a specific food or type of food. Recently, research has shown that mindfulness practices are effective in reducing negative emotions and the intensity of food cravings. Particularly, the body scan meditation has been shown to reduce rumination, improve emotion regulation, decrease negative affect and increase positive affect. However, no research so far has examined the effects of the body scan meditation on the intensity of food cravings through the reduction of the negative emotions that elicit the craving. Given the empirically supported ability of the body scan meditation to facilitate changes in the perceived body boundaries and spatial frames of reference and to consequently reduce negative emotions, the investigators can expect that reduced body boundaries and a more allocentric frame of reference will mediate the ability of the body scan meditation to reduce negative affect and cravings. Finding such effects through the hypothesized mechanisms would contribute to the knowledge on how mindfulness-based exercises exert their positive influence. Furthermore, if the body scan is found to be an effective means of reducing negative affect and consequently the intensity of food cravings, it could be recommended to emotional eaters as one practice to regulate their emotions and eating behaviors.

Thus, the current study will use a pre-post randomized-controlled study to examine whether the body scan reduces induced negative affect and food cravings in emotional eaters through reduced salience of body boundaries and a more allocentric spatial frame of reference. The investigators predict that emotional eaters in the body scan condition will report more diffuse body boundaries, a more allocentric frame of reference, and lower rumination than emotional eaters in the control condition and that this will mediate reduced negative affect and, thereby, reduced cravings. Furthermore, the investigators predict that mindfulness, equanimity, cognitive defusion, and interoceptive awareness will act as moderators of the influence of the body scan meditation on negative affect and food cravings because individuals who score high on these variables will be more likely to benefit from the body scan meditation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who self-report as emotional eaters, indicated by a score of 3.25 or higher on the Dutch Eating Behavior Questionnaire (DEBQ; Van Strien et al., 1986)

Exclusion Criteria:

* Self-reported eating disorders
* Self-reported psychiatric conditions
* More than 10 hours of formal meditation practice (e.g., sitting meditation) or retreat experience in the last one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Negative affect subscale of the Positive and Negative Affect Scale | The investigators are assessing change from baseline (immediately after the mood induction) to immediately after the intervention.
  Negative affect will be measured using the negative affect subscale of the Positive and Negative Affect Scale. The lowest score is 10, and the highest score is 50. The higher outcome would mean a worse outcome as this indicates higher negative affect, and a lower score would indicate a better outcome (lower negative affect).
Desire subscale of the Food Cravings Questionnaire-State Version | The investigators are assessing change from baseline (immediately after the mood induction) to immediately after the intervention.
  The intensity of food cravings will be measured using the Desire subscale of Food Cravings Questionnaire- State Version. Three items that target cravings for food from the Desire subscale of Food Cravings Questionnaire- State Version will be used in the current study. Specifically, participants rate the three items: "I am craving tasty food", "I have an urge for tasty food", "I have an intense desire to eat tasty food." All items will be rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The mean score on the three items will be used as the food craving measure.

SECONDARY OUTCOMES:
Perceived Body Boundaries Scale | The investigators are assessing change from baseline (immediately after the mood induction) to immediately after the intervention
  Perceived body boundaries are described as the degree to which the self is experienced as a discrete, body-encapsulated entity, separate and isolated from the surrounding world. Participants are asked to rate the strength of their perceived body boundary between self and the world using a 7-point Likert type scale (1 = weak boundary, 7 = strong boundary). Scores are ranked from 0.0 to 15.5, and higher scores indicate higher salience in perceived body boundaries (better score), and lower scores indicate lower salience in perceived body boundaries (worse score).
Spatial Frame of Reference Continuum | Immediately after the mood induction and immediately after the intervention
  Spatial frame of reference is defined as the region within one's perception, often based in the body and construed as the self, that is involved in the sense of connection between self, others, and the environment
Brief State Rumination Inventory | Immediately after the mood induction and immediately after the intervention
  Rumination involves repetitively focusing attention on the causes and implications of one's negative mood.

OTHER OUTCOMES:
Adherence Checks | Immediately after the intervention
  The adherence checks will be adapted from the mind wandering check used in Dambrun et al. (2019). Participants will be asked two questions: to indicate the estimated percentage of time (from 0 to 100%) they were preoccupied by thoughts of the past or future; and to indicate the percentage of time (from 0 to 100%) they were able to follow the instructions of the practice recording.
Multidimensional Assessment of Interoceptive Awareness- 2 | Up to 2 days before testing
  The multidimensional assessment of interoceptive awareness-2 is a 32-item multidimensional measure that assesses key aspects of the mind-body interaction, namely, interoceptive awareness. Respondents indicate on a 6-point Likert-type scale (from 0 = never to 5 = always) how much each statement applies to them. The multidimensional assessment of interoceptive awareness-2 has eight scales: noticing of body sensations, not distracting from negative (e.g., painful) sensations, not worrying about uncomfortable sensations, sustaining attention to sensations, awareness of the link between sensations and emotions, regulating psychological distress via attention to sensations, active listening to the body for insight, and experiencing one's body as safe and trustworthy. A higher score would mean individuals have a higher level of interoceptive awareness (better score), and a lower score would mean individuals have a lower level of interoceptive awareness (worse score).
Equanimity Scale | Up to 2 days before testing
  Equanimity is defined as an even-minded mental disposition towards all objects of experience regardless of their affective valence or source. This scale is to measure equanimity and contains 12 items assess the "even-minded state of mind," and the other 13 items measure "hedonic independence". The participants will use a 5-point Likert scale (1 = never or very rarely to 5 = very often or always) for this scale. A higher score would mean an individual has a more even-minded mental disposition towards all objects of experience (better score) and a lower score would mean an individual has less even-minded mental disposition towards all objects of experience (worse score)
Drexel Defusion Scale | Up to 2 days before testing
  Cognitive defusion is defined as the ability to gain psychological distance from thoughts and feelings by seeing them as mere events in the mind. Participants are asked to indicate the degree to which they would be able to defuse from hypothetical situations with negative thoughts or feelings on a 6-point Likert scale ranging from "not at all" (0) to "very much" (5). A higher score would indicate a greater ability to defuse from negative thoughts and feelings (better) and a lower score would indicate an individual is less able to defuse from negative thoughts and feelings (worse)
Five Factor Mindfulness Questionnaire | Up to 2 days before testing
  The five factor mindfulness questionnaire is a 39-item questionnaire in which respondents indicate on a 5-point Likert-type scale (from 1 = never or very rarely true to 5 = often or always true) how much various statements describe them. This questionnaire aims measures five facets of habitual or trait mindfulness: Observing, Describing, Acting with Awareness, Non-Judging of Internal Experiences, and Non-Reactivity to Inner Experiences ("I perceive my feelings and emotions without having to react to them"). A higher score would indicate a greater score of trait mindfulness, indicating greater ability to observe, describe, act with awareness, be non-judgmental of internal experiences, and non-reactive to inner experiences. A lower score indicates a lower level of all these indices (a worse score).

CONTACTS AND LOCATIONS:
Overall Officials: Huma Shireen, MA, MPsy, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annesi JJ, Johnson PH, Tennant GA, Porter KJ, Mcewen KL. Weight Loss and the Prevention of Weight Regain: Evaluation of a Treatment Model of Exercise Self-Regulation Generalizing to Controlled Eating. Perm J. 2016 Summer;20(3):15-146. doi: 10.7812/TPP/15-146. Epub 2016 Feb 1. PMID 26901268
- [Background] Ricca V, Castellini G, Fioravanti G, Lo Sauro C, Rotella F, Ravaldi C, Lazzeretti L, Faravelli C. Emotional eating in anorexia nervosa and bulimia nervosa. Compr Psychiatry. 2012 Apr;53(3):245-51. doi: 10.1016/j.comppsych.2011.04.062. Epub 2011 May 26. PMID 21620387
- [Background] Farb NA, Segal ZV, Mayberg H, Bean J, McKeon D, Fatima Z, Anderson AK. Attending to the present: mindfulness meditation reveals distinct neural modes of self-reference. Soc Cogn Affect Neurosci. 2007 Dec;2(4):313-22. doi: 10.1093/scan/nsm030. PMID 18985137
- [Background] Dambrun M. When the dissolution of perceived body boundaries elicits happiness: The effect of selflessness induced by a body scan meditation. Conscious Cogn. 2016 Nov;46:89-98. doi: 10.1016/j.concog.2016.09.013. Epub 2016 Sep 28. PMID 27684609
- [Background] Christoff K, Cosmelli D, Legrand D, Thompson E. Specifying the self for cognitive neuroscience. Trends Cogn Sci. 2011 Mar;15(3):104-12. doi: 10.1016/j.tics.2011.01.001. Epub 2011 Feb 1. PMID 21288760
- [Background] Hanley M, Khairat M, Taylor K, Wilson R, Cole-Fletcher R, Riby DM. Classroom displays-Attraction or distraction? Evidence of impact on attention and learning from children with and without autism. Dev Psychol. 2017 Jul;53(7):1265-1275. doi: 10.1037/dev0000271. Epub 2017 May 4. PMID 28471220
- [Background] Forman EM, Shaw JA, Goetter EM, Herbert JD, Park JA, Yuen EK. Long-term follow-up of a randomized controlled trial comparing acceptance and commitment therapy and standard cognitive behavior therapy for anxiety and depression. Behav Ther. 2012 Dec;43(4):801-11. doi: 10.1016/j.beth.2012.04.004. Epub 2012 Apr 24. PMID 23046782
- [Background] Desbordes G, Gard T, Hoge EA, Holzel BK, Kerr C, Lazar SW, Olendzki A, Vago DR. Moving beyond Mindfulness: Defining Equanimity as an Outcome Measure in Meditation and Contemplative Research. Mindfulness (N Y). 2014 Jan 21;2014(January):356-72. doi: 10.1007/s12671-013-0269-8. PMID 25750687
- [Background] Crosswell AD, Moreno PI, Raposa EB, Motivala SJ, Stanton AL, Ganz PA, Bower JE. Effects of mindfulness training on emotional and physiologic recovery from induced negative affect. Psychoneuroendocrinology. 2017 Dec;86:78-86. doi: 10.1016/j.psyneuen.2017.08.003. Epub 2017 Aug 4. PMID 28923751
- [Background] Forman EM, Herbert JD, Moitra E, Yeomans PD, Geller PA. A randomized controlled effectiveness trial of acceptance and commitment therapy and cognitive therapy for anxiety and depression. Behav Modif. 2007 Nov;31(6):772-99. doi: 10.1177/0145445507302202. PMID 17932235
- [Background] Sevinc G, Holzel BK, Hashmi J, Greenberg J, McCallister A, Treadway M, Schneider ML, Dusek JA, Carmody J, Lazar SW. Common and Dissociable Neural Activity After Mindfulness-Based Stress Reduction and Relaxation Response Programs. Psychosom Med. 2018 Jun;80(5):439-451. doi: 10.1097/PSY.0000000000000590. PMID 29642115
- [Background] Price CJ, Hooven C. Interoceptive Awareness Skills for Emotion Regulation: Theory and Approach of Mindful Awareness in Body-Oriented Therapy (MABT). Front Psychol. 2018 May 28;9:798. doi: 10.3389/fpsyg.2018.00798. eCollection 2018. PMID 29892247
- [Background] Gallagher S. Philosophical conceptions of the self: implications for cognitive science. Trends Cogn Sci. 2000 Jan;4(1):14-21. doi: 10.1016/s1364-6613(99)01417-5. PMID 10637618
- [Background] Jhangiani R, Tarry H, Stangor C. Principles of social psychology; 1st international edition.
- [Background] Deng Y-Q, Li S, Tang Y-Y. The relationship between wandering mind, depression and mindfulness. Mindfulness 2014;5(2):124-128.
- [Background] Hanley AW, Dambrun M, Garland EL. Effects of Mindfulness Meditation on Self-Transcendent States: Perceived Body Boundaries and Spatial Frames of Reference. Mindfulness (N Y). 2020 May;11(5):1194-1203. doi: 10.1007/s12671-020-01330-9. Epub 2020 Feb 14. PMID 33747250
- [Background] Austin JH. Zen-brain reflections. MIT press; 2010.
- [Background] Yaden DB, Haidt J, Hood RW, Vago DR, Newberg, AB. The varieties of self-transcendent experience. Review of General Psychology. 2017;21(2):143-160.
- [Background] Kabat-Zinn, Jon. Wherever You Go, There You Are: Mindfulness Meditation in Everyday Life. Hachette Books; 1994:104.
- [Background] Gendall KA, Joyce PR, Sullivan PF. Impact of definition on prevalence of food cravings in a random sample of young women. Appetite. 1997 Feb;28(1):63-72. doi: 10.1006/appe.1996.0060. PMID 9134095
- [Background] Dambrun M, Berniard A, Didelot T, Chaulet M, Sylvie DV, Corman M, Juneau C, Lea MM. Unified consciousness and the effect of body scan meditation on happiness: alteration of inner-body experience and feeling of harmony as central processes. Mindfulness. 2019;10(8):1530-1544.
- [Background] Dahl CJ, Lutz A, Davidson RJ. Reconstructing and deconstructing the self: cognitive mechanisms in meditation practice. Trends Cogn Sci. 2015 Sep;19(9):515-23. doi: 10.1016/j.tics.2015.07.001. Epub 2015 Jul 28. PMID 26231761
- [Background] Alberts HJ, Mulkens S, Smeets M, Thewissen R. Coping with food cravings. Investigating the potential of a mindfulness-based intervention. Appetite. 2010 Aug;55(1):160-3. doi: 10.1016/j.appet.2010.05.044. Epub 2010 May 21. PMID 20493913
- [Background] Alberts HJ, Thewissen R, Raes L. Dealing with problematic eating behaviour. The effects of a mindfulness-based intervention on eating behaviour, food cravings, dichotomous thinking and body image concern. Appetite. 2012 Jun;58(3):847-51. doi: 10.1016/j.appet.2012.01.009. Epub 2012 Jan 10. PMID 22265753
- [Background] Ng HH, Wu CW, Huang FY, Cheng YT, Guu SF, Huang CM, Hsu CF, Chao YP, Jung TP, Chuang CH. Mindfulness Training Associated With Resting-State Electroencephalograms Dynamics in Novice Practitioners via Mindful Breathing and Body-Scan. Front Psychol. 2021 Oct 28;12:748584. doi: 10.3389/fpsyg.2021.748584. eCollection 2021. PMID 34777144
- [Background] Frayn M, Knäuper B. Emotional eating and weight in adults. Current Psychology: A Journal for Diverse Perspectives on Diverse Psychological Issues. 2018; 37(4):924-933.
- [Background] Hanley AW, Garland EL. Spatial frame of reference as a phenomenological feature of self-transcendence: Measurement and manipulation through mindfulness meditation. Psychology of Consciousness: Theory, Research, and Practice. 2019; 6(4): 329-345.
- [Background] Sauer-Zavala SE, Walsh EC, Eisenlohr-Moul TA, Lykins, EB. Comparing mindfulness-based intervention strategies: Differential effects of sitting meditation, body scan, and mindful yoga. Mindfulness. 2013; 4(4): 383-388.
- [Background] James W. The self. The self in social interaction. 1968;141-49.